CLINICAL TRIAL: NCT02361645
Title: Vitreous Nonsteroidal Antiinflammatory Drus Concentrations And Prostaglandin E2 Levels in Vitrectomy Patients Treated With Indomethacin 0.5%, Bromfenac 0.09%, and Nepafenac 0.1%
Brief Title: NSAIDs and PGE2 Levels in Vitrectomy Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Russo, PhD Candidate, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vitreo001
Record Dates: First submitted 2015-01-27; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Vitreous Inflammation
Keywords: nonsteroidal antiinflammatory drugs; prostaglandin E2; vitrectomy
MeSH Terms: interventions — Ketorolac; Ophthalmic Solutions; Indomethacin; bromfenac; nepafenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control Group (No Intervention): No NSAIDs were administered prior to surgery
- Ketorolac eyedrops (Experimental): Ketorolac 0.5% eyedrops were administered prior to surgery
  Interventions: Drug: Ketorolac 0.5% eyedrops
- Indomethacin eyedrops (Experimental): Indomethacin 0.5% eyedrops were administered prior to surgery
  Interventions: Drug: Indomethacin 0.5% eyedrops
- Nepafenac eyedrops (Experimental): Nepafenac 0.1% eyedrops were administered prior to surgery
  Interventions: Drug: Nepafenac 0.1% eyedrops
- Bromfenac eyedrops (Experimental): Bromfenac 0.09% eyedrops were administered prior to surgery
  Interventions: Drug: Bromfenac 0.09% eyedrops

INTERVENTIONS:
Drug: Ketorolac 0.5% eyedrops
  Arms: Ketorolac eyedrops
Drug: Indomethacin 0.5% eyedrops
  Arms: Indomethacin eyedrops
Drug: Bromfenac 0.09% eyedrops
  Arms: Bromfenac eyedrops
Drug: Nepafenac 0.1% eyedrops
  Arms: Nepafenac eyedrops

SUMMARY:
The purpose of this study is to assess vitreous concentrations of nonsteroidal antiinflammatory drugs (NSAIDs) and prostaglandin E2 in patients treated with NSAIDs before vitrectomy.

A total of 0.5 to 1 mL undiluted vitreous was removed from the midvitreous cavity at the beginning of the surgery before infusion with balanced salt solution. Samples were immediately frozen and stored at -40°C until analysis. Samples were evaluated in a masked fashion. Vitreous concentrations of the study drugs were quantified using a reverse-phase liquid chromatography mass spectroscopy system. The minimum quantification limit for ketorolac, bromfenac, nepafenac, and amfenac was 0.8 ng/mL. Prostaglandin E2 concentrations were determined using a commercially available competitive enzyme immunoassay kit (R & D Systems, Minneapolis, MN).

ELIGIBILITY:
Inclusion Criteria:

* patients with pucker scheduled for vitrectomy

Exclusion Criteria:

* diabetes
* active inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Prostaglandin E2 levels in the vitreous (pg/mL) | 7 days after NSAID TID administration, following vitrectomy

SECONDARY OUTCOMES:
NSAIDs concentration (ng/mL) into the vitreous | 7 days after NSAID TID administration, following vitrectomy
  Vitreous concentrations of the study drugs were quantified using a reverse phase high performance liquid chromatography mass spectroscopy system.
Adverse events | 7 days after NSAID TID administration, following vitrectomy

REFERENCES:
- [Derived] Morescalchi F, Russo A, Semeraro F. SURGICAL OUTCOMES OF VITREOMACULAR TRACTION TREATED WITH FOVEAL-SPARING PEELING OF THE INTERNAL LIMITING MEMBRANE. Retina. 2021 Oct 1;41(10):2026-2034. doi: 10.1097/IAE.0000000000003139. PMID 33595256